CLINICAL TRIAL: NCT01986465
Title: Comparing the Effectiveness of Steroid Injection Versus Placebo and Immobilization Versus no Immobilization in Treating Patients With Lateral Epicondylitis
Brief Title: Effectiveness of Steroid Injection in Treating Patients With Lateral Epicondylitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amir Moayednia, Dr., Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 387278
Record Dates: First submitted 2013-11-11; First posted 2013-11-18 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-11

CONDITIONS: Lateral Epicondylitis
Keywords: lateral epicondylitis; treatment; steroid; immobilization
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Depomedrol (Experimental): The trial pharmacist prepares a series of similar vials containing either 4 mg of Depomedrol or Normal Saline and coded them either 1, 2, 3 or 4, the group assignments are not decoded until the end of the trial when the final analysis is due to take place. Patients take their envelopes to the trial pharmacist who give them a coded vial which they take to the orthopaedic surgeon who make the injection. After the injection the trial clerk take the patients to a technician who give patients in groups 1 and 3 long arm splints.
  Interventions: Drug: Depomedrol
- Placebo (Placebo Comparator): The trial pharmacist prepares a series of similar vials containing either 4 mg of Depomedrol or Normal Saline and coded them either 1, 2, 3 or 4, the group assignments are not decoded until the end of the trial when the final analysis is due to take place. Patients take their envelopes to the trial pharmacist who give them a coded vial which they take to the orthopaedic surgeon who make the injection. After the injection the trial clerk take the patients to a technician who give patients in groups 1 and 3 long arm splints.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Depomedrol
  Arms: Depomedrol
Drug: Placebo
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate the effectiveness of steroid injection and immobilization versus no immobilization in treating patients with lateral epicondylitis.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 65 years
* confirmed lateral epicondylitis
* had not received any treatment prior to enrolment

Exclusion Criteria:

* symptoms lasting less than 6 weeks
* history of acute trauma, fracture, and/or surgery within 12 months
* patients who had received corticosteroid injection, physiotherapy, splint or casting during the past 6 months
* bilateral involvement and history of cervical disk herniation, radiculopathy or abnormal electrophysiologic study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2013-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Function | Within the first 24 weeks after therapy
  The trial subjects are evaluated using the Oxford Elbow Scale (OES). They are asked to come to the trial office at 2 weeks, 4 weeks and 24 weeks for follow-up evaluation by administration of OES.
Pain | Within the first 24 weeks after therapy
  The trial subjects are evaluated using the Oxford Elbow Scale (OES). They are asked to come to the trial office at 2 weeks, 4 weeks and 24 weeks for follow-up evaluation by administration of OES.
Social-psychological | Within the first 24 weeks after therapy
  The trial subjects are evaluated using the Oxford Elbow Scale (OES). They are asked to come to the trial office at 2 weeks, 4 weeks and 24 weeks for follow-up evaluation by administration of OES.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad A Tahririan, MD, Principal Investigator — Isfahan University of Medical Sciences
Locations (1):
- Kashani University Hospital, Isfahan, Isfahan, Iran

REFERENCES:
- [Background] Ahmad Z, Siddiqui N, Malik SS, Abdus-Samee M, Tytherleigh-Strong G, Rushton N. Lateral epicondylitis: a review of pathology and management. Bone Joint J. 2013 Sep;95-B(9):1158-64. doi: 10.1302/0301-620X.95B9.29285. PMID 23997125